CLINICAL TRIAL: NCT07143617
Title: Exploratory Clinical Study on the Safety of STR-P004 in the Treatment of Patients With Relapsed or Refractory Autoimmune Diseases
Brief Title: Exploratory Clinical Study on the Safety of STR-P004
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing GoBroad Hospital (Other)
Collaborators: Starna Therapeutics (Industry)
Responsible Party: Principal Investigator, Jing Pan, Principal Investigator, Beijing GoBroad Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BJGBYY-IIT-LCYJ-2025-063
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Autoimmune Diseases
Keywords: STR-P004; Autoimmune Diseases; in-vivo Cart
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DL-1 STR-P004 Amg/kg (Experimental): Enrolled patients will receive Amg/kg of STR-P004 Intravenous infusion
  Interventions: Biological: STR-P004
- DL1 STR-P004 Bmg/kg (Experimental): Enrolled patients will receive Bmg/kg of STR-P004 Intravenous infusion
  Interventions: Biological: STR-P004
- DL2 STR-P004 Cmg/kg (Experimental): Enrolled patients will receive Cmg/kg of STR-P004 Intravenous infusion
  Interventions: Biological: STR-P004

INTERVENTIONS:
Biological: STR-P004 — STR-P004 Intravenous infusion

SUMMARY:
This is an open-label, multiple-dose escalation IIT clinical study aimed at evaluating the safety, tolerability, PK, and preliminary efficacy of STR-P004 in adult patients with relapsed or refractory autoimmune diseases.

DETAILED DESCRIPTION:
This study adopts the "TITE-BOIN12" dose escalation method and plans to set 3 dose groups: DL-1 Amg/kg, DL1 Bmg/kg, DL2 Cmg/kg, where DL-1 is a backup dose reduction group, and the starting dose group is DL1. If one or more DLTs occur in the first 3 subjects enrolled in DL1, the study will fallback to the backup dose reduction group and implement the TITE-BOIN12 dose escalation and expansion strategy starting from the DL-1 dose group. This study will only make dose escalation and OBD selection decisions based on the safety and efficacy data of SLE-ITP subjects. Subjects with other indications will only be enrolled at the confirmed safe dose level of the SLE-ITP cohort (i.e., based on the DLT rate of the current dose group, the dose adjustment decision is not to reduce the dose) and will not participate in dose escalation and OBD selection decisions.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand the purpose, nature, method of the trial and possible adverse reactions, voluntarily participate as a subject, and sign the informed consent form.
2. Aged ≥18 years (including the boundary value, based on the time of signing the informed consent form), male or female;
3. Applicable to Systemic Lupus Erythematosus (SLE):

   1. Diagnosed with Systemic Lupus Erythematosus (SLE) according to the 2019 European League Against Rheumatism (EULAR)/1997 American College of Rheumatology (ACR) classification criteria for diagnosis.
   2. SLE-ITP: platelet count < 50×10^9/L in at least 2 consecutive blood routine tests; no obvious abnormalities in blood cell morphology by peripheral blood smear microscopy; bone marrow cell morphology consistent with immune thrombocytopenia; excluding thrombocytopenia caused by other non-SLE reasons, such as infection, bone marrow suppression, splenomegaly, hypersplenism, etc.; failed to achieve at least partial response after receiving at least 1 course of MP pulse therapy (1g×3 days) or high-dose hormone (1mg/kg/d equivalent glucocorticoid) combined with 1 or more immunosuppressants. Note: Complete Response (CR): platelet count ≥100×10^9/L; Partial Response (PR): platelet count 30-100×10^9/L, at least twice the pre-treatment level, and no bleeding.
4. Other SLE: despite standard treatment, SLEDAI-2000 score ≥8 points and at least one BILAG Grade A or two BILAG Grade B; meeting one of the following conditions: positive antinuclear antibody (ANA) confirmed during screening, or anti-dsDNA antibody higher than normal level at screening, or anti-Sm antibody higher than normal level at screening; before the first administration of the trial drug, the subject has received at least one of the following standard treatments for 12 weeks, and the dose must be stable (dose reduction is allowed, dose increase is not allowed) for at least 30 days. Standard treatment regimens refer to stable use of any of the following: a. Antimalarial drugs combined with oral glucocorticoids (OCS, such as prednisone or equivalent dose of other hormones) and/or immunosuppressants (including mycophenolate mofetil, cyclophosphamide, leflunomide, methotrexate, tacrolimus, cyclosporine, azathioprine, tripterygium wilfordii); b. OCS and/or immunosuppressant combination therapy. If the subject is receiving OCS (such as prednisone or equivalent dose of other hormones), the following conditions must be met: the maximum dose of OCS at screening and during screening is 30 mg/day prednisone (or equivalent dose of other hormones); other drugs and traditional Chinese medicines that affect immunity can be continued at the discretion of the investigator; Applicable to Idiopathic Inflammatory Myopathies (IIM):

   1. Diagnosed with possible or definite Idiopathic Inflammatory Myopathies (IIM) according to the 2017 European League Against Rheumatism (EULAR)/American College of Rheumatology (ACR) classification criteria for diagnosis -- possible IIM: score of 5.5 points without biopsy; definite IIM: score of 6.7 points with biopsy; meeting the definition of refractory or relapsed IIM;
   2. Definition of refractory IIM: receiving at least one immunosuppressant (such as azathioprine, methotrexate, mycophenolate mofetil, cyclosporine, tacrolimus, cyclophosphamide, leflunomide, etc.) at a stable dose for more than 2 months, and when glucocorticoids are reduced to 10mg prednisone per day or equivalent dose or higher, at least one of the following deteriorations occurs: (i) progression of ILD, worsening of exertional dyspnea, or increase in ILD score on lung HRCT, or decrease in FVC% predicted value of pulmonary function by more than 5%, or decrease in DLco% by >10%; (ii) worsening of myositis, decrease in MMT-8 by >5 points/150 points, or increase in creatine kinase by >100U/L compared with previous levels;
   3. Definition of relapsed IIM: recurrence of active IIM causing new organ involvement or aggravation of originally involved organs after 6 months of continuous remission, or requiring an increase in glucocorticoids and immunosuppressants.

Exclusion Criteria:

1. Severe lupus nephritis within 8 weeks before screening (defined as urinary protein >6 g/24 hours or serum creatinine >2.5 mg/dL or 221 μmol/L), or need to use protocol-prohibited drugs to treat active nephritis, or need hemodialysis or receive prednisone ≥100 mg/d or equivalent glucocorticoid treatment for ≥14 days;
2. Central nervous system diseases caused by SLE or non-SLE within 8 weeks before screening (including but not limited to epilepsy, psychosis, interstitial encephalopathy syndrome, cerebrovascular accident, encephalitis, central nervous system vasculitis, etc.);
3. Other types of idiopathic inflammatory myopathies: inclusion body myositis, atrophic diabetes, juvenile myositis; patients with severe muscle damage or myositis with permanent weakness or cardiac involvement caused by non-IIM reasons (such as stroke);
4. SSc-related pulmonary hypertension requiring treatment; or rapidly progressive SSc-related lower gastrointestinal tract (small and large intestine) involvement (requiring parenteral nutrition), active gastric antral vascular ectasia; previous renal crisis caused by SSc;
5. History of important organ transplantation (such as heart, lung, kidney, liver) or hematopoietic stem cell/bone marrow transplantation;
6. Concurrent with two or more immune diseases requiring systemic treatment, which the investigator deems unsuitable for enrollment;
7. Suffering from IgA deficiency (serum IgA level <10 mg/dL);
8. Participation in any other clinical trial within 4 weeks before screening or within 5 half-lives of the trial drug (whichever is longer);
9. Previous receipt of CAR-T therapy or other cell or gene therapy;
10. Receipt of belimumab within 2 weeks before screening; receipt of B cell-depleting drugs such as rituximab or equivalent therapy (targeting CD19, CD20, BAFF, etc.) within 1 month before screening, unless it can be proven that B cells have recovered to pre-treatment levels or within the normal range;
11. Receipt of anti-SLE treatment other than standard treatment (such as Saphnelo) within 3 months before screening or within 5 half-lives of the drug (whichever is longer);
12. Receipt of live/attenuated vaccine within 4 weeks before screening or planned to receive live/attenuated vaccine during the trial;
13. Uncontrolled active infection;
14. Admission or evidence of use of illicit drugs, drug abuse, or alcoholism;
15. Receipt of major surgery within 4 weeks before screening or minor surgery within 2 weeks before screening; wounds must be completely healed (surgical procedures such as catheter placement are not exclusion criteria);
16. History of any of the following cardiovascular diseases within 6 months before screening: New York Heart Association (NYHA) class III or IV heart failure, myocardial infarction, unstable angina pectoris, uncontrolled or symptomatic atrial arrhythmia, any ventricular arrhythmia, or other heart diseases with significant clinical significance;
17. Any other severe underlying diseases (such as active gastric ulcer, uncontrolled epileptic seizures, cerebrovascular events, gastrointestinal bleeding, severe signs and symptoms of coagulation and coagulation dysfunction, heart disease), mental diseases, psychological, familial, or regional diseases that the investigator determines may interfere with planned staging, treatment, and follow-up, affect patient compliance, or put the patient at high risk of complications;
18. Evidence of concurrent malignant tumors within <5 years before screening, except for fully treated cervical carcinoma in situ, localized cutaneous squamous cell carcinoma, basal cell carcinoma, localized prostate cancer, breast ductal carcinoma in situ, or ≤T1 urothelial carcinoma. Patients with prostate cancer under active surveillance are eligible to participate in this study;
19. Pregnant or lactating women;
20. Viral serological test during screening: positive for human immunodeficiency virus antibody (HIV-Ab); positive for hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibody (HBc-Ab), and HBV-DNA copy number greater than the measurable lower limit; positive for hepatitis C antibody (HCV-Ab) and HCV-RNA copy number greater than the measurable lower limit; or subjects with positive treponema pallidum antibody (TP-Ab);
21. Subjects with active or latent tuberculosis (positive T-SPOT) detected during screening;
22. Receipt of splenectomy for treatment within 6 months before screening;
23. Other subjects deemed unsuitable for participation in this trial by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-09-14 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT), all adverse events (AEs)/serious adverse events (SAEs); | 12 months

IPD SHARING:
Plan to Share IPD: No